CLINICAL TRIAL: NCT03421392
Title: Study of Platelets Sialylation by Flow Cytometry for the Differential Diagnosis of Immunologic and Constitutive Thrombocytopenia: Diagnostic and Prognostic Interest.
Brief Title: Study of Platelets Sialylation by Flow Cytometry for the Differential Diagnosis of ICT
Acronym: SYMPATHIC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0346
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: constitutive thrombocytopenia; central thrombocytopenia; platelets; sialylation; flow cytometry
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Idiopathic thrombocytopenic purpura
  Interventions: Other: non interventional study
- non immunological thrombocytopenia: patient with constitutive thrombocytopenia, myelodysplastic syndrome, or chemotherapy-induced thrombocytopenia
  Interventions: Other: non interventional study
- without thrombocytopenia
  Interventions: Other: non interventional study

INTERVENTIONS:
Other: non interventional study — non interventional study

SUMMARY:
Idiopathic thrombocytopenic purpura (ITP) is the most frequent auto-immune cytopenia. There is no specific biological marker and the diagnosis often results from the exclusion of other differential diagnoses, notably inherited thrombocytopenia.

Recent studies have reported an original platelet destruction mechanism in ITP, by antibody-mediated desialylation of membrane proteins. The detection of platelet sialylation can be readily achieved using flow cytometry. This could provide a new biomarker of ITP, useful to ascertain a diagnosis of ITP and guide towards proper patient management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18yo) with a diagnosis of ITP (primary acute, persisting or chronical)
* Adult patients (>18yo) with a diagnosis of non immunological thrombocytopenia (constitutive thrombocytopenia, myelodysplastic syndrome, chemotherapy-induced thrombocytopenia)
* Adult patients (>18 yo) without thrombocytopenia
* Enrolled in a Social Security system
* Having provided informed consent

Exclusion Criteria:

* Minor patients (<18 yo)
* Enrolled in another clinical study
* Having received corticosteroids or polyvalent immunoglobulins in the past 4
* weeks or anti-platelet therapy or NSAID during the past 7 days
* Having received platelet transfusion in the past fortnight
* With proven iron deficiency
* With drug-induced immune-allergic thrombocytopenia.
* Pregnant and breastfeeding women,
* guardian patients, will be excluded from this population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 Populations will be recruited in the study:
  Number of topics planned:
  50 Patients in the PTI group 50 patients in the non-immunological thrombocytopenia group 50 patients in the control group
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Assess the difference of sialylation between ITP patients and other causes of thrombocytopenia / controls | 18 months
  a significant decrease in platelets sialylation in ITP patients, measured in flow cytometry with fluorescent Ricinus communis agglutinin

SECONDARY OUTCOMES:
Prognostic value and therapy | 18 months
  prognostic value of the level of sialylation in ITP patients regarding disease evolution and response of first line treatments and splenectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fouassier, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, van der Wal DE, Zhu G, Xu M, Yougbare I, Ma L, Vadasz B, Carrim N, Grozovsky R, Ruan M, Zhu L, Zeng Q, Tao L, Zhai ZM, Peng J, Hou M, Leytin V, Freedman J, Hoffmeister KM, Ni H. Desialylation is a mechanism of Fc-independent platelet clearance and a therapeutic target in immune thrombocytopenia. Nat Commun. 2015 Jul 17;6:7737. doi: 10.1038/ncomms8737. PMID 26185093
- [Background] Sorensen AL, Rumjantseva V, Nayeb-Hashemi S, Clausen H, Hartwig JH, Wandall HH, Hoffmeister KM. Role of sialic acid for platelet life span: exposure of beta-galactose results in the rapid clearance of platelets from the circulation by asialoglycoprotein receptor-expressing liver macrophages and hepatocytes. Blood. 2009 Aug 20;114(8):1645-54. doi: 10.1182/blood-2009-01-199414. Epub 2009 Jun 11. PMID 19520807